CLINICAL TRIAL: NCT03368911
Title: The Effect of Reinforced Endotracheal Tube on Post-operative Hoarseness
Brief Title: The Effect of Reinforced Endotracheal Tube on Post-operative Hoarseness Undergoing Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Seongtae Jeong, Associate Professor, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CNUHH-2017-102
Record Dates: First submitted 2017-11-30; First posted 2017-12-11 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Voice Hoarseness; Sore Throat; Thyroidectomy
Keywords: Hoarseness; Sore Throat; Thyroidectomy
MeSH Terms: conditions — Hoarseness; Pharyngitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Primary outcome is assessed by other investigator who do not know which endotrachdeal tube is used.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reinforced tube group (Experimental): use an reinforced endotracheal tube for endotracheal intubation during general anesthesia undergoing thyroidectomy
  Interventions: Device: Oral/Nasal Endotracheal Tube, Reinforced (Covidien)
- Conventional tube group (Active Comparator): use an conventional endotracheal tube for endotracheal intubation during general anesthesia undergoing thyroidectomy
  Interventions: Device: TaperGuard oral tracheal tube (Covidien)

INTERVENTIONS:
Device: Oral/Nasal Endotracheal Tube, Reinforced (Covidien) — Use Oral/Nasal Endotracheal Tube, Reinforced (Covidien) for endotracheal intubation
  Arms: Reinforced tube group
Device: TaperGuard oral tracheal tube (Covidien) — Use TaperGuard oral tracheal tube (Covidien) for endotracheal intubation
  Arms: Conventional tube group

SUMMARY:
The purpose of this study is an evaluation of the effect of the reinforced endotracheal tube on post-operative hoarseness and sore throat undergoing thyroidectomy

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist physical status 1-3
* Patients undergoing thyroidectomy under general anesthesia
* Tumor size < 2cm
* Patient who do not have any problem in the vocal cord

Exclusion Criteria:

* Patient who is expected difficult intubation (Mallampati class 3 or more)
* Patient who has respiratory disorder
* Previous hoarseness and sore throat history
* Obesity (BMI > 30 kg/m2)
* Recurrent laryngeal injury during operation
* Operation history of oral and laryngeal surgery

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
hoarseness | assess after 1hours after operation
  compare the incidence and degree of the hoarseness after thyroidectomy
sore throat | assess after 1hours after operation
  compare the incidence and degree of the sore throat after thyroidectomy
hoarseness | assess after 24 hours after operation
  compare the incidence and degree of the hoarseness after thyroidectomy
sore throat | assess after 24hours after operation
  compare the incidence and degree of the sore throat after thyroidectomy
hoarseness | assess after 48 hours after operation
  compare the incidence and degree of the hoarseness after thyroidectomy
sore throat | assess after 48 hours after operation
  compare the incidence and degree of the sore throat after thyroidectomy

CONTACTS AND LOCATIONS:
Overall Officials: Seongtae Jeong, Principal Investigator — Chonnam National University Hospital
Locations (2):
- South Korea (2):
  - Chonnam National University Hwasun Hopspital, Hwasun, Jeollanamdo
  - Chonnam National University Hospital, Gwangju

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR